CLINICAL TRIAL: NCT00040261
Title: An Investigation of the Antidepressant Efficacy of Memantine, an NMDA Antagonist With Neurotrophic Properties in Major Depression
Brief Title: Clinical Trial of Memantine for Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020231; 02-M-0231
Record Dates: First submitted 2002-06-22; First posted 2002-06-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Depression
Keywords: Antiglutamatergic; Neuroprotective; Unipolar Depression; Treatment; Antidepressant; Depression; Glutamate; Memantine; Pathophysiology; Positron Emission Tomography; Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major | interventions — Memantine

INTERVENTIONS:
Drug: Memantine HCL

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the drug memantine for treating major depression.

Major depression is a serious public health concern that contributes to significant morbidity and mortality. Despite the availability of a wide range of antidepressant drugs, a proportion of patients with major depression fail to respond to first-line antidepressant treatment, despite adequate dosage, duration, and compliance. Recent studies suggest that the glutamatergic system may play a role in the pathophysiology and treatment of depression. Memantine and other agents which reduce glutamatergic neurotransmission may represent a novel class of antidepressants.

The study consists of three phases. In Phase 1, participants will be tapered off all psychiatric medications over a 2-week washout period. In Phase 2, participants will be randomly assigned to receive either memantine or placebo (an inactive pill) three times a day for 8 weeks. Participants who do not respond to the treatment after 8 weeks will be taken off the study and offered standard treatment. Weekly psychiatric evaluations will evaluate treatment response. During Phase 2, participants who respond well to treatment will enter Phase 3, a 16-week continuation phase of either memantine or placebo. Interviews will be conducted every other week in the first month , then monthly thereafter.

Participants will have a physical examination, neuropsychological tests, and eye blink tests at baseline and at the end of the study. Pulse, blood pressure, and blood samples will be taken throughout the study. Participants will undergo an electrocardiogram as well as positron emission tomography (PET) and magnetic resonance imaging (MRI) scans of the brain.

DETAILED DESCRIPTION:
Major affective disorders are common, severe, chronic and often a life-threatening illness. Major depression contributes to significant morbidity and mortality. Impairment in physical and social functioning resulting from depression can be just as severe as other chronic medical illnesses. Suicide is the cause of death in 10-20% of individuals with recurrent depressive disorders.

Despite the availability of a wide range of antidepressant drugs, clinical trials indicate that 30% to 40% of patients with major depression fail to respond to first-line antidepressant treatment, despite adequate dosage, duration, and compliance. Thus, there is a clear need to develop novel and improved therapeutics for unipolar and bipolar depression. Recent preclinical studies suggest that antidepressants may exert delayed indirect effects on the glutamatergic system. Furthermore, a growing body of data suggests that mood disorders are associated with regional volumetric reductions, and cell loss and atrophy. It is thus noteworthy that lamotrigine, which, among other effects reduces glutamate release, has antidepressant effects, and a pilot study has suggested that NMDA antagonists may have antidepressant effects. Together, this data suggests that the glutamatergic system may play a role in the pathophysiology and treatment of depression, and that agents, which more directly reduce glutamatergic neurotransmission, may represent a novel class of antidepressants.

Memantine (Akatinol memantine), an agent that is approved in Germany for dementia syndrome, Parkinson's disease has significant antiglutamatergic and neuroprotective properties, may prove to have antidepressant properties in depressed patients. In this study, we propose to investigate the potential efficacy of memantine, an agent which reduces glutamatergic output via open-channel block of the NMDA receptor-associated ion channel. Most importantly, memantine only blocks the channel during periods of abnormal, excessive activity, and leaves relatively spared normal neurotransmission. This finding is the basis for the minimal side effect profile displayed by memantine.

Patients, ages 18 to 80, with a diagnosis of major depression (without psychotic features), will be randomized to double-blind treatment outpatient study to receive either memantine (5-20mg/day) or placebo for a period of 8 weeks. Following this acute period, patients who fully respond could enter a 16-week continuation phase. Acute efficacy will be determined by demonstrating a greater response rate using specified criteria. Approximately 112 patients with acute major depression will be enrolled in the study.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects may be included in the study only if they meet all of the following criteria:

Male or female subjects, 18 to 80 years of age.

Female subjects of childbearing potential must be using a medically accepted means of contraception.

Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol.

Subjects must be considered reliable.

Each subject must understand the nature of the study and must sign an informed consent document.

Subjects must fulfill the criteria for major depression, recurrent without psychotic features as defined in DSM-IV based on clinical assessment and confirmed by structured diagnostic interview SCID-P.

Subjects must have an initial score at Visit 1 and Visit 2 of at least 22 on the MADRS.

Subjects must not have a decrease in the total score of MADRS of greater than 20 % during washout (between Visits 1 and 2).

Current major depressive episode of at least 4 weeks duration.

EXCLUSION CRITERIA:

Subjects will be excluded from the study for any of the following reasons:

Lack of response to more than 2 antidepressants (adequate dose and duration).

Participation in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry (Visit 1).

Female subjects who are either pregnant or nursing.

Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

Subjects with uncorrected hypothyroidism or hyperthyroidism.

Subjects with one or more seizures without a clear and resolved etiology.

Documented history of hypersensitivity or intolerance to amantadine or prior treatment with memantine.

DSM-IV substance abuse or dependence (except nicotine and caffeine) within the past 90 days.

Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to Visit 2.

Treatment with a reversible monoamine oxidase inhibitor, guanethidine, or guanadrel within 1 week prior to Visit 2.

Treatment with fluoxetine within 6 weeks prior to Visit 2.

Treatment with any other concomitant medication with primarily CNS activity.

Treatment with clozapine within 4 weeks prior to Visit 2.

Treatment with amitriptyline (elavil) within 4 weeks prior to Visit 2 since amitriptyline and similar TCAs may manifest a mild NMDA receptor antagonism, as demonstrated in electrophysiological studies.

Treatment with the anticonvulsants carbamazepine (tegretol, carbatrol, tegretol XR and similar derivatives), gabapentin (neurontin) or felbamate (felbatol) within 4 weeks prior to Visit 2 because these drugs may interfere with NMDA receptor function.

Treatment with electroconvulsive therapy (ECT) within 3 months (90 days) prior to Visit 2.

Current diagnosis of schizophrenia or other psychotic or bipolar disorder as defined in the DSM-IV.

Judged clinically to be at serious suicidal risk.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112
Dates: Start 2002-06; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Altamura CA, Mauri MC, Ferrara A, Moro AR, D'Andrea G, Zamberlan F. Plasma and platelet excitatory amino acids in psychiatric disorders. Am J Psychiatry. 1993 Nov;150(11):1731-3. doi: 10.1176/ajp.150.11.1731. PMID 8214185
- [Background] Auer DP, Putz B, Kraft E, Lipinski B, Schill J, Holsboer F. Reduced glutamate in the anterior cingulate cortex in depression: an in vivo proton magnetic resonance spectroscopy study. Biol Psychiatry. 2000 Feb 15;47(4):305-13. doi: 10.1016/s0006-3223(99)00159-6. PMID 10686265
- [Background] Ambrozi L, Danielczyk W. Treatment of impaired cerebral function in psychogeriatric patients with memantine--results of a phase II double-blind study. Pharmacopsychiatry. 1988 May;21(3):144-6. doi: 10.1055/s-2007-1014666. PMID 3406051
- [Derived] Lepow L, Luckenbaugh DA, Park L, Henter ID, Zarate CA Jr. Case series: Antidepressant effects of low-affinity and low-trapping NMDA receptor antagonists did not predict response to ketamine in seven subjects. J Psychiatr Res. 2017 Mar;86:55-57. doi: 10.1016/j.jpsychires.2016.10.023. Epub 2016 Nov 22. No abstract available. PMID 27914292